CLINICAL TRIAL: NCT01931956
Title: A Continued Access Registry of the Evalve® MitraClip® System: EVEREST II Real World Expanded Multicenter Study of the MitraClip System (REALISM)
Brief Title: Real World Expanded Multicenter Study of the MitraClip® System (REALISM)
Acronym: REALISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0401B; 0401 (Other: Abbott Vascular)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency
Keywords: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Mitral Valve Incompetence; Mitral Regurgitation; Mitral Insufficiency; Mitral Valve; Mitral Regurgitation (MR); Mitral Valve Prolapse; Edge to Edge (E2E); Alfieri Technique; MitraClip; Functional MR; Degenerative MR; Echocardiogram; Coronary Artery Disease (CAD); Heart Failure; Heart Attack; EVEREST; EVEREST I; EVEREST II; REALISM
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Coronary Artery Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Non-High Risk (Experimental): Includes patients who are candidate for mitral valve repair or replacement surgery, including cardiopulmonary bypass (i.e. non-high risk). The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant. This arm was evaluated as a separate study NCT00209274.
  Interventions: Device: MitraClip® implant
- High Risk (Experimental): Includes patients with a predicted procedural mortality risk calculated using the Society For Thoracic Surgeon (STS) surgical risk calculator of ≥12% or, in the judgment of a cardiac surgeon, the patient is considered a high risk surgical candidate due to the presence of pre-defined risk factors. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant. This arm was evaluated as a separate study NCT01940120.
  Interventions: Device: MitraClip® implant
- Compassionate Use (Experimental): Patients that did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either Emergency Use (EU) or Compassionate Use (CU). The objective of the Compassionate and Emergency Use Group of the EVEREST II REALISM study is to provide access to the MitraClip Device, in a non-commercial setting, for patients with serious or life-threatening conditions when conventional therapies have failed, are unsuitable, or unavailable. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
  Interventions: Device: MitraClip® implant
- Emergency Use (Experimental): Patients that did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either Emergency Use (EU) or Compassionate Use (CU). The objective of the Compassionate and Emergency Use Group of the EVEREST II REALISM study is to provide access to the MitraClip Device, in a non-commercial setting, for patients with serious or life-threatening conditions when conventional therapies have failed, are unsuitable, or unavailable. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
  Interventions: Device: MitraClip® implant

INTERVENTIONS:
Device: MitraClip® implant — Percutaneous mitral valve repair using MitraClip implant

SUMMARY:
Prospective, multicenter, continued access registry of the MitraClip® Cardiovascular Valve Repair System in the treatment of mitral valve regurgitation. Patients will undergo 30-day, 6-month, 12-month, 36-month and 60-month clinical follow-up. The study consists of two arms: a High Risk group (NCT01940120) and a Non-High Risk group (NCT00209274) . Patients that did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either Emergency Use (EU) or Compassionate Use (CU).

DETAILED DESCRIPTION:
The EVEREST II REALISM study (REALISM study) is a continued access registry designed for continued data collection on the use of Abbott Vascular's MitraClip System (MitraClip® Device) under more "real world" conditions. After the completion of enrollment in the pivotal EVEREST II Randomized Controlled Trial (RCT) NCT00209274 and EVEREST II High Risk Registry Study NCT01940120, continued access to the technology was warranted to collect additional safety and effectiveness data on the MitraClip® Device. This continued access study was approved by FDA on November 21, 2008 (G030064). There are two arms (High Risk and Non-High Risk) in the REALISM study. Patients that did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either Emergency Use (EU) or Compassionate Use (CU). Enrollment in the Non-High Risk arm of the study concluded on April 14, 2011 and enrollment in the High Risk arm concluded on December 19, 2013.

REALISM is a prospective, multi-center, study of the safety and effectiveness of an endovascular approach to the treatment of mitral valve regurgitation using the Evalve Cardiovascular Valve Repair System (MitraClip® implant). Patients with moderate-to-severe (3+) or severe (4+) mitral regurgitation (MR), as determined by the site from a transthoracic echocardiogram (TTE), were considered for enrollment in this study. The TTE and a transesophageal echocardiogram (TEE) are used to assess eligibility criteria for MR severity, valve anatomy and left ventricular parameters.

ELIGIBILITY:
Patients screened in EVEREST II REALISM Study will first be screened for high risk (HR) status and enrolled into the HR arm if they meet eligibility for this arm of the study. If they do not meet eligibility for the HR arm, patients will be further screened for eligibility for enrollment into the non-high risk (NHR) arm.

Key Inclusion Criteria:

* The primary regurgitant jet originates from malcoaptation of the A2 and P2 scallops of the mitral valve (MV)
* Male or non-pregnant female
* Trans-septal catheterization is determined to be feasible by the treating physician

High Risk Arm:

* Predicted procedural mortality risk calculated using the STS surgical risk calculator of ≥12% or, in the judgment of a cardiac surgeon, the patient is considered a HR surgical candidate due to the presence of one of the following indications:

  1. Porcelain aorta or mobile ascending aortic atheroma
  2. Post-radiation mediastinum
  3. Previous mediastinitis
  4. Functional MR with EF <40
  5. Over 75 years old with EF<40
  6. Re-operation with patent grafts
  7. Two or more prior chest surgeries
  8. Hepatic cirrhosis
  9. Three or more of the following STS high risk factors 9.1 Creatinine >2.5 mg/dL 9.2 Prior chest surgery 9.3 Age over 75 9.4 EF<35
* Symptomatic moderate to severe (3+) or severe (4+) chronic MR and in the judgment of the investigator intervention to reduce MR is likely to provide symptomatic relief for the patient
* American Society of Anesthesiologists (ASA) physical status classification of ASA IV or lower

Non-High Risk Arm:

* Moderate to severe (3+) or severe (4+) chronic MV regurgitation and:

  1. Symptomatic with >25% LVEF and LVESD ≤55mm or, 2. Asymptomatic with one or more of the following: i. Left Ventricular Ejection Fraction (LVEF) 25% to 60% ii. Left Ventricular End-Systolic Diameter (LVESD) ≥40 mm iii. New onset of Atrial fibrillation (AFib) iv. Pulmonary arterial systolic pressure (PASP) >50 mmHg at rest or >60 mmHg with exercise
* Candidate for MV repair or replacement surgery, including cardiopulmonary bypass

Key Exclusion Criteria:

* Evidence of an Acute Myocardial Infarction (AMI) in the prior 12 weeks of the intended treatment
* In the judgment of the Investigator, the femoral vein cannot accommodate a 24 French scale (F) catheter or the presence of an inferior vena cava (IVC) filter would interfere with advancement of the catheter or ipsilateral Deep Venous Thrombus (DVT) is present
* MV orifice area <4.0 cm2
* If leaflet flail is present:

  1. Flail Width ≥15 mm, or
  2. Flail Gap ≥10 mm.
* If leaflet tethering is present:

  1. Vertical coaptation length <2 mm
* Leaflet anatomy which may preclude clip implantation, proper clip positioning on the leaflets or sufficient reduction in MR. This may include:

  1. Evidence of calcification in the grasping area of the A2 and/or P2 scallops
  2. Presence of a significant cleft of A2 or P2 scallops
  3. More than one anatomic criteria dimensionally near the exclusion limits
  4. Bileaflet flail or severe bileaflet prolapse
  5. Lack of both primary and secondary chordal support
* Hemodynamic instability (systolic pressure <90 mmHg without afterload reduction or cardiogenic shock or the need for inotropic support or intra-aortic balloon pump).
* Need for emergency surgery for any reason
* Prior MV surgery or valvuloplasty or any currently implanted mechanical prosthetic valve or currently implanted Ventricular assist device (VAD)
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* Active endocarditis or active rheumatic heart disease or leaflets degenerated from either endocarditis or rheumatic disease (i.e. noncompliant, perforated)
* History of bleeding diathesis or coagulopathy or subject will refuse blood transfusions
* Life expectancy <12 months
* Active infections requiring current antibiotic therapy
* Patients in whom transesophageal echocardiography (TEE) is contraindicated

High Risk Arm:

* EF <20%, and/or LVESD >60 mm

Non-High Risk Arm:

* The need for any other cardiac surgery
* Any endovascular therapeutic interventional or surgical procedure performed within 30 days prior to the index procedure
* Severe Left Ventricular (LV) dysfunction (EF <25% and/or LVESD >55mm)
* Severe mitral annular calcification
* Systolic anterior motion of the MV leaflet
* Hypertrophic cardiomyopathy
* History of a stroke or documented Transient Ischemic Attack (TIA) within the prior 6 months
* Upper GI bleeding within the prior 6 months
* Platelet count <75,000 cells/mm³
* Creatinine >2.5mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 965 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted Feldman, M.D. Feldman, M.D., Study Director — Endeavor Health; Donald D Glower Jr., MD, Study Director — Duke University
Locations (38):
- United States (38):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Hospital of Miami, FL, Miami, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - The Care Group Medical Center (St. Vincent Hospital), Indianapolis, Indiana
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Terrebonne General Medical Center, Houma, Louisiana
  - Maine Medical Center, Portland, Maine
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - St. Patrick's Hospital & Health Science Center, Missoula, Montana
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York University Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Carolina's Medical Center (Sanger Clinic), Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina Heart Institute, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Grayburn PA, Roberts BJ, Aston S, Anwar A, Hebeler RF Jr, Brown DL, Mack MJ. Mechanism and severity of mitral regurgitation by transesophageal echocardiography in patients referred for percutaneous valve repair. Am J Cardiol. 2011 Sep 15;108(6):882-7. doi: 10.1016/j.amjcard.2011.05.013. Epub 2011 Jul 7. PMID 21741608
- [Result] Pope NH, Lim S, Ailawadi G. Late calcific mitral stenosis after MitraClip procedure in a dialysis-dependent patient. Ann Thorac Surg. 2013 May;95(5):e113-4. doi: 10.1016/j.athoracsur.2012.10.067. PMID 23608290
- [Result] Glower DD, Kar S, Trento A, Lim DS, Bajwa T, Quesada R, Whitlow PL, Rinaldi MJ, Grayburn P, Mack MJ, Mauri L, McCarthy PM, Feldman T. Percutaneous mitral valve repair for mitral regurgitation in high-risk patients: results of the EVEREST II study. J Am Coll Cardiol. 2014 Jul 15;64(2):172-81. doi: 10.1016/j.jacc.2013.12.062. PMID 25011722
- [Derived] Ailawadi G, Lim DS, Mack MJ, Trento A, Kar S, Grayburn PA, Glower DD, Wang A, Foster E, Qasim A, Weissman NJ, Ellis J, Crosson L, Fan F, Kron IL, Pearson PJ, Feldman T; EVEREST II Investigators. One-Year Outcomes After MitraClip for Functional Mitral Regurgitation. Circulation. 2019 Jan 2;139(1):37-47. doi: 10.1161/CIRCULATIONAHA.117.031733. PMID 30586701
- [Derived] Wang A, Sangli C, Lim S, Ailawadi G, Kar S, Herrmann HC, Grayburn P, Foster E, Weissman NJ, Glower D, Feldman T. Evaluation of renal function before and after percutaneous mitral valve repair. Circ Cardiovasc Interv. 2015 Jan;8(1):e001349. doi: 10.1161/CIRCINTERVENTIONS.113.001349. PMID 25593120
- [Derived] Lim DS, Reynolds MR, Feldman T, Kar S, Herrmann HC, Wang A, Whitlow PL, Gray WA, Grayburn P, Mack MJ, Glower DD. Improved functional status and quality of life in prohibitive surgical risk patients with degenerative mitral regurgitation after transcatheter mitral valve repair. J Am Coll Cardiol. 2014 Jul 15;64(2):182-92. doi: 10.1016/j.jacc.2013.10.021. Epub 2013 Oct 31. PMID 24184254
- See also: Web site listing study sites and describing mitral regurgitation, symptoms, clinical consequences and treatments — https://www.vascular.abbott/us/homepage.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of February 13, 2018, a total of 59 Compassionate Use and 7 Emergency Use patients have undergone MitraClip procedure between 14 Dec 2010 and 22 Feb 2013. A total of 628 patients in the High Risk arm between January 22, 2009 and December 19, 2013 and 271 patients in the Non-High Risk arm were enrolled between January 22, 2009 and April 14, 2011.
Pre-assignment Details: Patients who did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either EU or CU.
Groups:
- Emergency Use: Patients that did not meet REALISM High Risk or Non-High Risk eligibility criteria were evaluated for consideration for either Emergency Use (EU) or Compassionate Use (CU). The objective of the Compassionate and Emergency Use Group of the EVEREST II REALISM study is to provide access to the MitraClip Device, in a non-commercial setting, for patients with serious or life-threatening conditions when conventional therapies have failed, are unsuitable, or unavailable. All EU patients had a medical condition that in the opinion of the investigators was likely to result in death within 30 days. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
- High Risk: Includes patients with a predicted procedural mortality risk calculated using the Society For Thoracic Surgeon (STS) surgical risk calculator of ≥12% or, in the judgment of a cardiac surgeon, the patient is considered a high risk surgical candidate due to the presence of pre-defined risk factors. The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
- Non-high Risk: Includes patients who are candidate for mitral valve repair or replacement surgery, including cardiopulmonary bypass (i.e. non-high risk).
  If a patient was not a candidate for the high risk arm, but met all other eligibility criteria for the non-high risk arm, the patient was enrolled into the non-high risk arm of EVEREST II REALISM.
  The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant
Period: Overall Study
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Started | 59 | 7 | 628 | 271
Completed | 8 | 0 | 141 | 138
Not Completed | 51 | 7 | 487 | 133
Not completed — Death | 42 | 7 | 379 | 96
Not completed — Withdrawal by Subject | 5 | 0 | 70 | 30
Not completed — Lost to Follow-up | 2 | 0 | 11 | 7
Not completed — Expected | 2 | 0 | 6 | 0
Not completed — Not due | 0 | 0 | 21 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk | Total
Number analyzed (Participants) | 59 | 7 | 628 | 271 | 965
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 75 | 41 | 125
  >=65 years | 51 | 6 | 553 | 230 | 840
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (9.2) | 78.6 (11.1) | 76.7 (10.7) | 73.9 (11.2) | 75.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 253 | 127 | 400
  Male | 42 | 4 | 375 | 144 | 565
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 34 | 9 | 46
  Not Hispanic or Latino | 56 | 7 | 594 | 262 | 919
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 1 | 0 | 8 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 47 | 12 | 63
  White | 54 | 6 | 563 | 246 | 869
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 9 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 59 | 7 | 628 | 271 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events
Description: A combined clinical endpoint of death, myocardial infarction (MI), re-operation for failed surgical repair or replacement, non-elective cardiovascular surgery for adverse events, stroke, renal failure, deep wound infection, ventilation for greater than 48 hours, gastro-intestinal (GI) complication requiring surgery, new onset of permanent atrial fibrillation, septicemia and transfusion of 2 or more units of blood.
Time Frame: 30 days
Population: Intent-To-Treat Population set (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- Non-high RIsk: Includes patients who are candidate for mitral valve repair or replacement surgery, including cardiopulmonary bypass (i.e. non-high risk).
  If a patient was not a candidate for the high risk arm, but met all other eligibility criteria for the non-high risk arm, the patient was enrolled into the non-high risk arm of EVEREST II REALISM The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high RIsk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 5 | 3 | 98 | 31

2. Primary Outcome: Number of Participants With Major Adverse Events
Description: A combined clinical endpoint of death, myocardial infarction (MI), re-operation for failed surgical repair or replacement, non-elective cardiovascular surgery for adverse events, stroke, renal failure, deep wound infection, ventilation for greater than 48 hours, GI complication requiring surgery, new onset of permanent atrial fibrillation, septicemia and transfusion of 2 or more units of blood.
Time Frame: 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- High Risk: Includes patients with a predicted procedural mortality risk calculated using the Society For Thoracic Surgeon (STS) surgical risk calculator of ≥12% or, in the judgment of a cardiac surgeon, the patient is considered a high risk surgical candidate due to the presence of pre-defined risk factors.
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 31 | 5 | 223 | 74

3. Primary Outcome: Number of Participants With 12-Month Efficacy
Description: Defined as freedom from: Surgery for Mitral Regurgitation (MR) or Valve Dysfunction, death, and MR > 2+ (moderate to severe (3+) or severe MR (4+)).
Time Frame: 12 months
Population: Analysis was performed in 52 participants out of 59 in CU arm, in 6 subjects out of 7 in EU arm, in 556 participants out of 628 participants and 248 out of 271 participants in non-HR arm were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 52 | 6 | 556 | 248
Participants | 25 | 1 | 339 | 166

4. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: The definition of a serious adverse event is an event that is fatal or life threatening, results in persistent or significant disability, requires intervention to prevent permanent impairment/damage, or an event that results in congenital anomaly, malignancy, hospital admission or prolongation of hospitalization.
Time Frame: 30 days
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
participants | 11 | 5 | 204 | 68

5. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: as for outcome 4
Time Frame: 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 37 | 7 | 388 | 131

6. Secondary Outcome: Number of Participants With Clinically Significant Atrial Septal Defect (ASD)
Description: Defined as a significant residual atrial septal opening. Reported as clinically significant if intervention is performed for the primary purpose of repairing the ASD. If cardiac surgery is indicated for reasons other than residual ASD (e.g., residual MR) and the ASD is repaired at the same time, this does not meet the definition of clinically significant ASD.
Time Frame: 30 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 2 | 0 | 14 | 11

7. Secondary Outcome: Number of Participants With Clinically Significant Atrial Septal Defect (ASD)
Description: as for outcome 6
Time Frame: 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- High Risk: Includes patients with a predicted procedural mortality risk calculated using the Society For Thoracic Surgeon (STS) surgical risk calculator of ≥12% or, in the judgment of a cardiac surgeon, the patient is considered a high risk surgical candidate due to the presence of pre-defined risk factors.The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
- Non-high Risk: Includes patients who are candidate for mitral valve repair or replacement surgery, including cardiopulmonary bypass (i.e. non-high risk).
  If a patient was not a candidate for the high risk arm, but met all other eligibility criteria for the non-high risk arm, the patient was enrolled into the non-high risk arm of EVEREST II REALISM.
  The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implants.
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 3 | 0 | 22 | 15

8. Secondary Outcome: Number of Participants With Major Adverse Events (MAE) in Patients Over 75 Years of Age
Description: MAE is defined as a combined clinical endpoint of Death (all cause), MI, Re-operation for Failed Surgical Repair or replacement, non-elective Cardiovascular Surgery for AEs, Stroke, Renal Failure, Deep Wound Infection, Ventilation for greater than 48 hours, GI complication requiring surgery, new onset of Permanent Afib, Septicemia, and transfusion of 2 or more units of blood. The occurrence of MAE is measured in patients over 75 years of age.
Time Frame: 30 days
Population: CU Arm:
  There are 27 patients >75 years old in the CU arm. Safety data are available only for 26 patients.
  EU Arm:
  There are 5 patients >75 years old in the EU arm.
  HR arm:
  There are 393 patients >75 years old in the HR arm.
  Non-HR arm:
  There are 140 patients >75 years old in the Non-HR arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 26 | 5 | 393 | 140
Participants | 3 | 2 | 64 | 16

9. Secondary Outcome: Number of Participants With Major Adverse Events in Patients Over 75 Years of Age
Description: as for outcome 8
Time Frame: 12 Months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 26 | 5 | 393 | 140
Participants | 14 | 3 | 139 | 40

10. Secondary Outcome: Number of Participants With Major Adverse Events in Patients Over 75 Years of Age
Description: as for outcome 8
Time Frame: 2 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 26 | 5 | 393 | 140
Participants | 14 | 4 | 146 | 40

11. Secondary Outcome: Number of Participants With Major Adverse Events in Patients Over 75 Years of Age
Description: as for outcome 8
Time Frame: 3 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 26 | 5 | 393 | 140
Participants | 14 | 4 | 146 | 40

12. Secondary Outcome: Number of Participants With Major Adverse Events in Patients Over 75 Years of Age
Description: as for outcome 8
Time Frame: 4 years
Population: CU Arm:
  There are 27 patients >75 years old in the CU arm. Safety data are available only for 24 patients.
  EU Arm:
  There are 5 patients >75 years old in the EU arm.
  HR arm:
  There are 393 patients >75 years old in the HR arm.
  Non-HR arm:
  There are 140 patients >75 years old in the Non-HR arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 24 | 5 | 393 | 140
Participants | 12 | 4 | 146 | 40

13. Secondary Outcome: Number of Participants With Major Adverse Events in Patients Over 75 Years of Age
Description: as for outcome 8
Time Frame: 5 years
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 24 | 5 | 393 | 140
Participants | 12 | 4 | 146 | 40

14. Secondary Outcome: Number of Participants With Acute Procedural Success
Description: Defined as successful implantation of the Clip(s) with resulting MR severity of 2+ or less as determined by the echocardiographic assessment at discharge. The 30-day echocardiogram will be used if the discharge echocardiogram is unavailable or uninterpretable, providing the patient has not undergone subsequent surgery after attempted clip.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 41 | 3 | 524 | 229

15. Secondary Outcome: Number of Participants With Procedural Success
Description: Defined as successful implantation of the Clip(s) with resulting MR severity of 2+ of less at discharge or a 1 grade MR reduction at discharge accompanied by a 1 level reduction in NYHA at 30 days.
Time Frame: 30 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 45 | 4 | 541 | 239

16. Secondary Outcome: Number of Participants With Clinical Durability
Description: Defined as the proportion of patients who have an acute reduction in MR severity of at least one grade (as measured by the discharge echocardiogram) that at 12 months have not required surgery for valve dysfunction and meet either of the following: 1) MR severity grade of 2+ or less or 2) a one grade reduction in MR severity compared to baseline accompanied by at least a one level reduction in NYHA at 12 months.
Time Frame: 12 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 22 | 0 | 325 | 163

17. Secondary Outcome: Number of Participants With Clip Implant Rate
Description: Defined as the procedural rate of successful delivery and deployment of Clip implants with echocardiographic evidence of leaflet approximation and retrieval of the investigational delivery catheter.
Time Frame: On the day of index procedure (≤1 day)
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Non-high Risk: Includes patients who are candidate for mitral valve repair or replacement surgery, including cardiopulmonary bypass (i.e. non-high risk). If a patient was not a candidate for the high risk arm, but met all other eligibility criteria for the non-high risk arm, the patient was enrolled into the nonhigh risk arm of EVEREST II REALISM The patients who are enrolled in this arm will undergo percutaneous mitral valve repair using MitraClip® implant.
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 55 | 7 | 603 | 258

18. Secondary Outcome: Procedure Time
Description: The mean procedure time is defined as the start time of the transseptal procedure to the time the steerable guide catheter (SGC) is removed.
Time Frame: On the day of index procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 58 | 7 | 619 | 262
minutes | 141.7 (70.4) | 123.6 (55.9) | 139.0 (66.8) | 137.8 (68.4)

19. Secondary Outcome: Device Time
Description: Device time is defined as the time of insertion of the Steerable Guide Catheter (SGC) to the time the MitraClip delivery catheter is retracted into the SGC.
Time Frame: On the day of index procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 58 | 7 | 616 | 262
minutes | 115.1 (65.6) | 96.6 (60.2) | 106.8 (58.2) | 111.5 (63.8)

20. Secondary Outcome: Fluoroscopy Duration
Description: Mean fluoroscopy duration during the MitraClip procedure.
Time Frame: On the day of index procedure
Population: ITT population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 627 | 269
minutes | 42.5 (28.9) | 33.6 (21.3) | 38.5 (24.4) | 34.6 (20.0)

21. Secondary Outcome: Number of Participants With MitraClip Devices Implanted
Description: The distribution of number of MitraClip devices implanted in patients.
Time Frame: On the day of index procedure
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants
  0 Clips | 4 | 0 | 25 | 13
  1 Clip | 30 | 5 | 333 | 160
  2 Clips | 25 | 2 | 268 | 98
  3 Clips | 0 | 0 | 2 | 0

22. Secondary Outcome: Post-Procedure Intensive Care Unit (ICU)/ Critical Care Unit (CCU)/ Post-anesthesia Care Unit (PACU) Duration
Description: Defined as the number of hours for which patients are in an intensive care unit or step down unit before discharge or moving to a standard care unit.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure).
Population: ITT population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 270
Hours | 22.1 (29.9) | 149.3 (179.3) | 36.5 (70.3) | 28.8 (69.5)

23. Secondary Outcome: Post-Procedure Length of Hospital Stay
Description: Defined as the number of days from the end of the procedure until the patient is discharged from the hospital. This does not include time in a nursing or skilled care facility.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure).
Population: ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 627 | 270
Days | 2.4 (2.4) | 12.3 (7.5) | 3.2 (4.6) | 2.8 (4.8)

24. Secondary Outcome: Number of Participants Experiencing Death
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: 12 months visit window (410 days)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 21 | 5 | 148 | 27
Participants
  Cardiac | 13 | 2 | 97 | 13
  Non-Cardiac | 7 | 3 | 49 | 14
  Not Adjudicated | 0 | 0 | 2 | 0
  Not Adjudicable | 1 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With Incidence of Discharge to a Nursing Home or Skilled Nursing Facility
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants
  Home | 51 | 0 | 523 | 248
  Home with home health care | 3 | 2 | 43 | 13
  Nursing home | 0 | 0 | 15 | 3
  Skilled nursing facility | 3 | 4 | 34 | 3
  Long-term acute care | 1 | 0 | 0 | 1
  Death | 1 | 1 | 12 | 2
  Withdrawal | 0 | 0 | 1 | 1

26. Secondary Outcome: Number of Participants With Hospital Re-admissions
Description: Defined as re-admission of patients to the hospital following discharge from the Clip procedure.
Time Frame: 30 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 7 | 1 | 74 | 15

27. Secondary Outcome: Number of Participants With Device Embolization or Single Leaflet Device Attachment (SLDA)
Description: A single leaflet device attachment (SLDA) is defined as attachment of one mitral valve leaflet to the MitraClip device.
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 0 | 1 | 13 | 11

28. Secondary Outcome: Number of Participants With Mitral Stenosis
Description: Mitral stenosis is a key safety consideration assessed after implantation of the MitraClip device. It is defined as Mitral Valve Area (MVA) less than 1.5 cm^2 as assessed by the Echocardiography Core Laboratory (ECL).
Time Frame: 0 to 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 55 | 7 | 603 | 258
Participants | 3 | 0 | 7 | 6

29. Secondary Outcome: Number of Participants With Mitral Regurgitation (MR) Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 30 days using echocardiography.
  MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 30 days(Follow-up)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 56 | 5 | 587 | 264
Participants
  0+: None | 0 | 0 | 7 | 1
  1+: Mild | 22 | 1 | 315 | 144
  2+: Moderate | 20 | 1 | 206 | 90
  3+: Moderate to Severe | 11 | 3 | 50 | 25
  4+: Severe | 3 | 0 | 9 | 4

30. Secondary Outcome: Number of Participants With MR Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 12 months using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 34 | 0 | 410 | 209
Participants
  0+: None | 1 | 0 | 6 | 3
  1+: Mild | 17 | 0 | 167 | 71
  2+: Moderate | 10 | 0 | 173 | 100
  3+: Moderate to Severe | 3 | 0 | 48 | 31
  4+: Severe | 3 | 0 | 16 | 4

31. Secondary Outcome: Number of Participants With MR Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 2 years using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 10 | 0 | 227 | 179
Participants
  0+: None | 0 | 0 | 0 | 4
  1+: Mild | 6 | 0 | 102 | 65
  2+: Moderate | 3 | 0 | 90 | 87
  3+: Moderate to Severe | 1 | 0 | 23 | 21
  4+: Severe | 0 | 0 | 12 | 2

32. Secondary Outcome: Number of Participants With MR Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 3 years using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 8 | 0 | 222 | 159
Participants
  0+: None | 1 | 0 | 1 | 8
  1+: Mild | 5 | 0 | 103 | 58
  2+: Moderate | 2 | 0 | 90 | 73
  3+: Moderate to Severe | 0 | 0 | 20 | 15
  4+: Severe | 0 | 0 | 8 | 5

33. Secondary Outcome: Number of Participants With MR Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 4 years using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 4 years
Population: The 4-year visit was optional and no data were collected at this time point for CU and EU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame in HR and Non-HR arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 66 | 67
Participants
  0+: None | 0 | 0 | 0 | 3
  1+: Mild | 0 | 0 | 29 | 26
  2+: Moderate | 0 | 0 | 32 | 22
  3+: Moderate to Severe | 0 | 0 | 4 | 14
  4+: Severe | 0 | 0 | 1 | 2

34. Secondary Outcome: Number of Participants With MR Severity
Description: Paired site-assessed Mitral regurgitation severity between baseline and 5 years using echocardiography. MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 5 | 0 | 108 | 117
Participants
  0+:None | 0 | 0 | 2 | 4
  1+:Mild | 4 | 0 | 50 | 50
  2+:Moderate | 1 | 0 | 43 | 48
  3+:Moderate to Severe | 0 | 0 | 10 | 9
  4+:Severe | 0 | 0 | 3 | 6

35. Secondary Outcome: Number of Participants With Second Intervention to Place an Additional Mitraclip Device.
Description: If residual MR was determined to be clinically unacceptable for patients who received only 1 clip during the index procedure, a second intervention to place an additional MitraClip device could be considered.
Time Frame: 139 days post the index procedure
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 1 | 0 | 12 | 3

36. Secondary Outcome: Number of Participants With Second Intervention to Place an Additional Mitraclip Device.
Description: as for outcome 35
Time Frame: 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 59 | 7 | 628 | 271
Participants | 1 | 0 | 33 | 11

37. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Functional Class
Description: Paired NYHA data from baseline to 30 days. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 50 | 3 | 560 | 252
Participants
  NYHA Functional Class I | 17 | 0 | 163 | 113
  NYHA Functional Class II | 22 | 2 | 296 | 110
  NYHA Functional Class III | 10 | 1 | 88 | 28
  NYHA Functional Class IV | 1 | 0 | 13 | 1

38. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: Paired NYHA data from baseline to 12 months. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 35 | 0 | 403 | 204
Participants
  NYHA Functional Class I | 14 | 0 | 157 | 121
  NYHA Functional Class II | 13 | 0 | 179 | 65
  NYHA Functional Class III | 7 | 0 | 61 | 18
  NYHA Functional Class IV | 1 | 0 | 6 | 0

39. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: Paired NYHA data from baseline to 2 years. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 23 | 0 | 293 | 182
Participants
  NYHA Functional Class I | 6 | 0 | 113 | 99
  NYHA Functional Class II | 11 | 0 | 126 | 68
  NYHA Functional Class III | 5 | 0 | 49 | 14
  NYHA Functional Class IV | 1 | 0 | 5 | 1

40. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: Paired NYHA data from baseline to 3 years. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 14 | 0 | 224 | 154
Participants
  NYHA Functional Class I | 7 | 0 | 82 | 85
  NYHA Functional Class II | 6 | 0 | 101 | 56
  NYHA Functional Class III | 1 | 0 | 34 | 12
  NYHA Functional Class IV | 0 | 0 | 7 | 1

41. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: Paired NYHA data from baseline to 4 years. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 4 years
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 105 | 125
Participants
  NYHA Functional Class I | 0 | 0 | 44 | 76
  NYHA Functional Class II | 0 | 0 | 47 | 35
  NYHA Functional Class III | 0 | 0 | 14 | 11
  NYHA Functional Class IV | 0 | 0 | 0 | 3

42. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: Paired NYHA data from baseline to 5 years. Class I: Patients with cardiac disease but without resulting limitations of physical activity.
  Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain.
  Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain.
  Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 6 | 0 | 121 | 119
Participants
  NYHA Functional Class I | 1 | 0 | 52 | 65
  NYHA Functional Class II | 3 | 0 | 48 | 49
  NYHA Functional Class III | 1 | 0 | 12 | 5
  NYHA Functional Class IV | 1 | 0 | 9 | 0

43. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 53 | 6 | 514 | 231
ml | 163.9 (68.2) | 110.7 (25.1) | 143.1 (54.1) | 121.8 (43.8)

44. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 0 | 335 | 179
ml | 171.1 (83.4) |  | 142.9 (57.3) | 120.9 (30.0)

45. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 190 | 153
ml | 175.0 (65.4) |  | 148.2 (68.2) | 119.6 (40.0)

46. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 195 | 141
ml | 155.7 (56.9) |  | 150.9 (69.0) | 120.1 (41.0)

47. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to 48 months as determined by the echo core laboratory.
Time Frame: 48 months
Population: For CU arm, there is no paired data available for 48 months as very few patients completed the 4 year follow-up and in EU arm all the patients died prior to 48 months. Thus the number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 54 | 63
ml |  |  | 138.6 (68.2) | 128.1 (38.2)

48. Secondary Outcome: Left Ventricular End-diastolic Volume (LVEDV)
Description: Paired Left ventricular end-diastolic volume (LVEDV) data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: For CU arm, there is no paired data available for 60 months as very few patients completed the 5 year follow-up and in EU arm all the patients died prior to 48 months. Thus the number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 97 | 100
ml |  |  | 146.1 (71.4) | 125.9 (45.6)

49. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 53 | 6 | 513 | 231
ml | 94.7 (58.9) | 46.3 (21.5) | 82.9 (44.7) | 59.4 (31.9)

50. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 0 | 354 | 179
ml | 102.2 (71.8) |  | 80.4 (48.6) | 57.6 (29.5)

51. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 189 | 153
ml | 98.7 (56.0) |  | 85.9 (59.0) | 57.1 (32.6)

52. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 194 | 141
ml | 97.0 (52.5) |  | 88.8 (60.2) | 55.8 (32.2)

53. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 54 | 63
ml |  |  | 77.8 (61.6) | 55.3 (26.5)

54. Secondary Outcome: Left Ventricular End-systolic Volume (LVESV)
Description: Paired Left ventricular end-systolic volume (LVESV) data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 97 | 100
ml |  |  | 85.4 (62.9) | 59.0 (38.2)

55. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 55 | 6 | 565 | 257
cm | 5.7 (1.2) | 4.6 (0.4) | 5.4 (0.8) | 5.1 (0.7)

56. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 34 | 0 | 396 | 201
cm | 5.9 (1.2) |  | 5.5 (0.9) | 5.1 (0.7)

57. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 9 | 0 | 213 | 169
cm | 5.9 (1.2) |  | 5.5 (1.0) | 5.0 (0.7)

58. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 8 | 0 | 215 | 156
cm | 5.9 (0.9) |  | 5.6 (1.0) | 5.2 (0.8)

59. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 61 | 68
cm |  |  | 5.5 (1.0) | 5.2 (0.7)

60. Secondary Outcome: Left Ventricular Internal Dimension Diastole (LVIDd)
Description: Paired Left Ventricular internal dimension diastole (LVIDd) data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 101 | 115
cm |  |  | 5.4 (1.0) | 5.3 (0.8)

61. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 55 | 6 | 542 | 242
cm | 4.5 (1.5) | 2.9 (0.5) | 4.3 (1.1) | 3.7 (0.8)

62. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 34 | 0 | 377 | 189
cm | 4.7 (1.5) |  | 4.2 (1.1) | 3.6 (0.9)

63. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 9 | 0 | 200 | 147
cm | 4.3 (1.6) |  | 4.3 (1.2) | 3.6 (0.9)

64. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 8 | 0 | 209 | 143
cm | 4.7 (1.3) |  | 4.4 (1.3) | 3.6 (1.0)

65. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 58 | 67
cm |  |  | 4.1 (1.4) | 3.6 (0.8)

66. Secondary Outcome: Left Ventricular Internal Dimension Systole (LVIDs)
Description: Paired Left Ventricular internal dimension systole (LVIDs) data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 101 | 110
cm |  |  | 4.2 (1.3) | 3.7 (1.0)

67. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 53 | 6 | 514 | 231
percentage of ejection fraction | 46.9 (15.5) | 59.4 (10.8) | 44.7 (13.1) | 53.0 (11.2)

68. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 0 | 355 | 179
percentage of ejection fraction | 46.0 (15.6) |  | 47.2 (14.0) | 53.9 (11.5)

69. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 190 | 153
percentage of ejection fraction | 47.0 (13.9) |  | 46.1 (14.2) | 54.4 (11.8)

70. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 194 | 141
percentage of ejection fraction | 41.5 (17.4) |  | 45.9 (15.0) | 55.5 (12.1)

71. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 54 | 63
percentage of ejection fraction |  |  | 48.9 (14.6) | 58.2 (8.5)

72. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Paired Left Ventricular Ejection Fraction (LVEF) data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 98 | 100
percentage of ejection fraction |  |  | 46.3 (14.6) | 55.5 (11.4)

73. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 50 | 6 | 479 | 216
cm | 4.1 (0.5) | 3.7 (0.5) | 3.8 (0.5) | 3.8 (0.5)

74. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 0 | 324 | 160
cm | 3.9 (0.4) |  | 3.8 (0.5) | 3.8 (0.5)

75. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 8 | 0 | 173 | 133
cm | 3.9 (0.2) |  | 3.8 (0.5) | 3.8 (0.5)

76. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 189 | 126
cm | 4.0 (0.3) |  | 3.9 (0.5) | 4.0 (0.5)

77. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 53 | 56
cm |  |  | 4.0 (0.5) | 4.1 (0.6)

78. Secondary Outcome: Septal-Lateral Annular Dimension Diastole (SLADd)
Description: Septal-Lateral Annular Dimension Diastole (SLADd) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in diastole. Paired SLADd data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 86 | 99
cm |  |  | 3.9 (0.5) | 4.0 (0.6)

79. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to discharge or 30 days as determined by echo core laboratory.
Time Frame: At discharge (an average of ≤ 12.3 days post-index procedure) or 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 50 | 6 | 472 | 212
cm | 3.5 (0.4) | 3.3 (0.6) | 3.4 (0.5) | 3.5 (0.4)

80. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to 12 months as determined by echo core laboratory.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 0 | 317 | 157
cm | 3.4 (0.4) |  | 3.3 (0.5) | 3.4 (0.5)

81. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to 24 months as determined by echo core laboratory.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 8 | 0 | 167 | 131
cm | 3.4 (0.3) |  | 3.3 (0.5) | 3.4 (0.5)

82. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to 36 months as determined by echo core laboratory.
Time Frame: 36 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 7 | 0 | 186 | 123
cm | 3.5 (0.4) |  | 3.4 (0.5) | 3.4 (0.5)

83. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to 48 months as determined by echo core laboratory.
Time Frame: 48 months
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 53 | 55
cm |  |  | 3.4 (0.5) | 3.5 (0.6)

84. Secondary Outcome: Septal-Lateral Annular Dimension Systole (SLADs)
Description: Septal-Lateral Annular Dimension systole (SLADs) is the dimension across the mitral valve from the anterior annulus to the posterior annulus at the widest point in the center of the valve, measured in systole.Paired SLADs data from baseline to 60 months as determined by echo core laboratory.
Time Frame: 60 months
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
Number analyzed (Participants) | 0 | 0 | 85 | 96
cm |  |  | 3.4 (0.6) | 3.5 (0.6)

85. Other Pre Specified Outcome: 36-Item Short Form Health Survey (SF-36) Quality of Life Change From Baseline to 30 Days
Description: The SF-36 is a multidimensional, patient-reported survey containing 36 questions on a 0-100 scale measuring physical (Physical Component Score PCS) & mental health status (Mental Component Score MCS) in relation to 8 health concepts:
  * Physical functioning
  * Role limitations due to physical or
  * Emotional health
  * Bodily pain
  * General health perceptions
  * Vitality
  * Social functioning
  * General mental health
  Responses to each of the SF-36 items are scored and expressed as a score on a 0-100 scale (0% in a domain represents the poorest possible QOL&100% indicates full QOL).Higher scores represent better self-perceived health.
  The physical & mental functions were assessed by the Physical Component Summary (PCS) score & Mental Component Summary (MCS) score. Normal PCS and MCS scores vary depending on the demographics of the population studied. The PCS&MCS norms for 65-75 year old are 44 & 52, respectively while the norms for CHF population are 31 & 46, respectively.
Time Frame: 30 days
Population: EU arm participants were not analyzed due to the serious/life-threatening conditions,SF-36 QOL data was not collected on all patients at baseline. Therefore, paired data at 30 days were not available for EU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Compassionate Use | High Risk | Non-high Risk
Number analyzed (Participants) | 44 | 500 | 93
Scores on a scale
  Physical Component Summary | 7.6 (9.6) | 38.3 (10.0) | 40.7 (9.6)
  Mental Component Summary | 5.3 (11.3) | 49.3 (12.0) | 52.5 (10.3)

86. Other Pre Specified Outcome: 36-Item Short Form Health Survey (SF-36) Quality of Life Change From Baseline to 12 Months
Description: as for outcome 85
Time Frame: 12 months
Population: EU arm participants were not analyzed due to the serious/life-threatening conditions, QOL data was not collected on all patients at baseline. Therefore, paired data at 1 year were not available for EU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Compassionate Use | High Risk | Non-high Risk
Number analyzed (Participants) | 32 | 332 | 77
Scores on a scale
  Physical Component Summary | 7.2 (10.7) | 38.9 (10.6) | 43.2 (10.6)
  Mental Component Summary | 6.7 (12.0) | 50.3 (11.9) | 51.3 (10.5)

87. Other Pre Specified Outcome: Change in 6-Minute Walk Test (6MWT)
Description: Defined as a cardiopulmonary function test that measures a patient's exercise capacity by the distance he or she can walk in six minutes.
Time Frame: At Baseline and 30 Days
Population: EU arm participants were not analyzed due to serious/life-threatening conditions, the 6MWT was not administered to all patients at baseline.Therefore,paired data at 30 days were not available for EU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame in CU, HR and Non-HR arms.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Compassionate Use | High Risk | Non-high Risk
Number analyzed (Participants) | 36 | 261 | 67
Meters
  Baseline | 243.1 (124.6) | 237.8 (141.9) | 386.7 (396.8)
  30 Days | 296.6 (186.8) | 278.8 (162.7) | 428.9 (296.4)
  Difference | 53.4 (131.4) | 40.9 (108.6) | 42.1 (293.5)

88. Other Pre Specified Outcome: Change in 6-Minute Walk Test (6MWT)
Description: as for outcome 87
Time Frame: At Baseline and 6 months
Population: EU and CU arm participants were not analyzed due to serious/life-threatening conditions, the 6MWT was not administered to all patients at baseline.Therefore, paired data at 6 months were not available for EU and CU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame HR and Non-HR arms.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | High Risk | Non-high Risk
Number analyzed (Participants) | 198 | 62
Meters
  Baseline | 252.0 (142.5) | 413.6 (406.4)
  6 Months | 283.8 (147.9) | 392.8 (245.1)
  Difference | 31.8 (134.7) | -20.9 (333.2)

89. Other Pre Specified Outcome: Change in 6-Minute Walk Test (6MWT)
Description: as for outcome 87
Time Frame: At Baseline and 12 months
Population: EU arm participants were not analyzed due to serious/life-threatening conditions, the 6MWT was not administered to all patients at baseline.Therefore, paired data at 1 year were not available for EU arm.
  The number of participants analyzed includes subjects who had available follow up data at that time frame in CU, HR and Non-HR arms.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Compassionate Use | High Risk | Non-high Risk
Number analyzed (Participants) | 25 | 172 | 57
Meters
  Baseline | 267.4 (115.3) | 261.4 (142.2) | 408.8 (380.3)
  12 Months | 291.4 (142.0) | 296.6 (129.9) | 392.6 (211.1)
  Difference | 24.0 (112.8) | 35.2 (155.7) | -16.2 (339.8)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Compassionate Use | Emergency Use | High Risk | Non-high Risk
All-Cause Mortality (participants affected / at risk) | 42/59 | 7/7 | 379/628 | 96/271
Serious Adverse Events (participants affected / at risk) | 49/59 | 7/7 | 542/628 | 208/271
Other Adverse Events (participants affected / at risk) | 39/59 | 4/7 | 503/628 | 225/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Compassionate Use (N=59) | Emergency Use (N=7) | High Risk (N=628) | Non-high Risk (N=271)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 49 | 23
Hematologic - Other (Blood and lymphatic system disorders) | 2 | 0 | 4 | 0
Infection (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Atrial arrhythmia (Cardiac disorders) | 4 | 1 | 43 | 35
Atrial septal defect (Cardiac disorders) | 1 | 0 | 9 | 2
Cardiac : other (Cardiac disorders) | 2 | 1 | 26 | 9
Cardiac arrest (Cardiac disorders) | 5 | 0 | 43 | 9
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 15 | 5
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 12 | 3
Chest pain (Cardiac disorders) | 2 | 0 | 31 | 11
Congestive heart failure (Cardiac disorders) | 13 | 3 | 232 | 63
Endocarditis (Cardiac disorders) | 1 | 0 | 5 | 4
Lead displacement (Cardiac disorders) | 1 | 0 | 1 | 1
Mitral stenosis (Cardiac disorders) | 1 | 0 | 4 | 2
Myocardial infarction (Cardiac disorders) | 4 | 0 | 26 | 7
Other rhythm disorder (Cardiac disorders) | 3 | 0 | 25 | 5
Residual/Recurrent MR (Cardiac disorders) | 3 | 1 | 35 | 26
Syncope/Dizziness (Cardiac disorders) | 1 | 0 | 24 | 5
Tamponade (Cardiac disorders) | 1 | 0 | 3 | 2
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 29 | 5
GI related - bleed (Gastrointestinal disorders) | 4 | 0 | 56 | 29
GI related - infection (Gastrointestinal disorders) | 2 | 0 | 9 | 7
GI related - other (Gastrointestinal disorders) | 7 | 2 | 65 | 23
Death (General disorders) | 34 | 7 | 352 | 95
Generalized weakness/fatigue (General disorders) | 1 | 0 | 20 | 6
Metabolic/endocrine disorders : Other (General disorders) | 1 | 0 | 41 | 24
Other (General disorders) | 7 | 0 | 73 | 34
device malfunction (General disorders) | 1 | 0 | 0 | 0
infection : Other (General disorders) | 2 | 0 | 23 | 10
Connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 | 0 | 57 | 30
Intracerebral hemorrhage (Nervous system disorders) | 1 | 0 | 15 | 3
Ischemic stroke (Nervous system disorders) | 1 | 0 | 3 | 4
Neurologic - other (Nervous system disorders) | 1 | 0 | 20 | 7
Stroke (Nervous system disorders) | 5 | 0 | 23 | 16
Mental disorders : Other (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal - infection (Renal and urinary disorders) | 1 | 0 | 20 | 9
Renal - other (Renal and urinary disorders) | 2 | 0 | 23 | 6
Renal - renal insufficiency/failure (Renal and urinary disorders) | 4 | 1 | 78 | 25
Bronchial/lung disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 23 | 6
Chronic obstructive pulmonary diseas (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 15 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 26 | 7
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 63 | 33
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 4
Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 46 | 18
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 56 | 26
Bleeding complication (Vascular disorders) | 2 | 0 | 32 | 10
Blood pressure complication (Vascular disorders) | 1 | 0 | 5 | 1
Deep vein thrombosis (DVT) (Vascular disorders) | 1 | 0 | 9 | 3
Embolization (Vascular disorders) | 2 | 0 | 2 | 1
Hematoma (Vascular disorders) | 1 | 0 | 12 | 6
Hemodynamic instability (Vascular disorders) | 2 | 1 | 28 | 6
Injury (Vascular disorders) | 1 | 0 | 1 | 1
Pseudoaneurysm (Vascular disorders) | 1 | 0 | 3 | 1
Vascular - other (Vascular disorders) | 1 | 0 | 12 | 9
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 12 | 5
Infection/bacteremia/septicemia (Blood and lymphatic system disorders) | 0 | 0 | 45 | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 6 | 4
Fever (General disorders) | 0 | 0 | 5 | 3
Skin/mucosal/subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8 | 5
AV fistula (Vascular disorders) | 0 | 0 | 1 | 2
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 3 | 2
Bruise/contusion/ecchymosis (Vascular disorders) | 0 | 0 | 1 | 0
Retroperitoneal hematoma (Vascular disorders) | 0 | 0 | 2 | 1
Stenosis (Vascular disorders) | 0 | 0 | 2 | 0
Transient Ischemic Attack (TIA) (Nervous system disorders) | 0 | 0 | 26 | 3
MV Surgery (Cardiac disorders) | 0 | 0 | 6 | 5
SLDA (Cardiac disorders) | 0 | 0 | 3 | 6
Coronary artery disease (Cardiac disorders) | 0 | 0 | 5 | 2
Heart transplant (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 3 | 1
Mitral valve injury (Cardiac disorders) | 0 | 0 | 3 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 4 | 5
peripheral edema (Cardiac disorders) | 0 | 0 | 6 | 1
Supraventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Thrombus (Cardiac disorders) | 0 | 0 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 7 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Bradyarrythmia (Cardiac disorders) | 0 | 0 | 10 | 4
Emergent MV surgery (Cardiac disorders) | 0 | 0 | 0 | 2
Hematologic-Shock (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Mesentric Ischemia (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Heart Block (Cardiac disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Compassionate Use (N=59) | Emergency Use (N=7) | High Risk (N=628) | Non-high Risk (N=271)
Anemia (Blood and lymphatic system disorders) | 5 | 1 | 69 | 32
Infection/Bacteremia/Septicemia (Blood and lymphatic system disorders) | 1 | 1 | 7 | 3
Other (Blood and lymphatic system disorders) | 1 | 0 | 8 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 22 | 10
Atrial Arrhythmia (Cardiac disorders) | 4 | 0 | 60 | 34
Atrial Septal Defect (Cardiac disorders) | 2 | 0 | 13 | 12
Bradyarrhythmia (Cardiac disorders) | 3 | 1 | 19 | 7
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 5 | 2
Chest Pain/Angina (Cardiac disorders) | 3 | 0 | 37 | 15
Congestive Heart Failure (Cardiac disorders) | 6 | 0 | 64 | 24
Lead Displacement (Cardiac disorders) | 1 | 0 | 2 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 22 | 6
Mitral Stenosis (Cardiac disorders) | 1 | 0 | 26 | 8
Mitral Valve Injury (Cardiac disorders) | 0 | 1 | 3 | 0
Other (Cardiac disorders) | 3 | 0 | 43 | 20
Other Rhythm Disorder (Cardiac disorders) | 4 | 0 | 24 | 12
Palpitations (Cardiac disorders) | 2 | 0 | 7 | 4
Pericardial Effusion (Cardiac disorders) | 2 | 0 | 8 | 16
Peripheral Edema (Cardiac disorders) | 3 | 1 | 33 | 18
Residual/Recurrent MR (Cardiac disorders) | 4 | 1 | 103 | 55
SLDA (Cardiac disorders) | 0 | 1 | 2 | 3
Syncope/Dizziness (Cardiac disorders) | 3 | 0 | 26 | 18
Thrombus (Cardiac disorders) | 1 | 0 | 4 | 1
Ventricular Arrhythmia (Cardiac disorders) | 2 | 0 | 17 | 6
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 21 | 5
Bleed (Gastrointestinal disorders) | 1 | 0 | 18 | 11
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 16 | 7
Other (Gastrointestinal disorders) | 3 | 2 | 85 | 44
Death (General disorders) | 1 | 0 | 3 | 0
Fever (General disorders) | 1 | 0 | 19 | 4
Generalized Weakness/Fatigue (General disorders) | 1 | 0 | 51 | 17
Infection (General disorders) | 4 | 0 | 18 | 7
Mental Disorders (General disorders) | 2 | 0 | 14 | 6
Metabolic/Endocrine Disorders (General disorders) | 5 | 0 | 70 | 35
Other (General disorders) | 7 | 1 | 141 | 62
Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 4 | 0 | 91 | 55
Confusion (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Nervous system disorders) | 0 | 1 | 0 | 0
Other (Nervous system disorders) | 5 | 2 | 53 | 15
Infection (Renal and urinary disorders) | 4 | 0 | 53 | 18
Other (Renal and urinary disorders) | 4 | 0 | 58 | 22
Renal Insufficiency/Failure (Renal and urinary disorders) | 8 | 0 | 66 | 26
Bronchial/Lung Disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 20 | 11
Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 20 | 11
Other (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 115 | 66
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 34 | 24
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 24 | 13
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 9 | 5
AV fistula (Vascular disorders) | 2 | 0 | 4 | 3
Aneurysm (Vascular disorders) | 1 | 0 | 4 | 1
Bleeding Complication (Vascular disorders) | 10 | 0 | 75 | 29
Blood Pressure Complication (Vascular disorders) | 2 | 0 | 15 | 12
DVT (Vascular disorders) | 1 | 0 | 6 | 2
Hematoma (Vascular disorders) | 4 | 0 | 55 | 15
Hemodynamic Instability (Vascular disorders) | 7 | 1 | 71 | 28
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 4 | 1
Endocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Heart block (Cardiac disorders) | 0 | 0 | 3 | 3
Myocardial infarction (Cardiac disorders) | 0 | 0 | 6 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 6 | 4
Supraventricular arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 3
Surgery (Cardiac disorders) | 0 | 0 | 1 | 0
Infection (Gastrointestinal disorders) | 0 | 0 | 9 | 6
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 8 | 3
Transient Ischemic Attack (TIA) (Nervous system disorders) | 0 | 0 | 13 | 9
Intracerebral hemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0
Ischemic stroke (Nervous system disorders) | 0 | 0 | 4 | 0
Stroke (Nervous system disorders) | 0 | 0 | 4 | 2
Incisional site pain (General disorders) | 0 | 0 | 20 | 13
Skin/mucosal/subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 0 | 11 | 8
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Peripheral Ischemia (Vascular disorders) | 0 | 0 | 2 | 1
Bruise/contusion/ecchymosis (Vascular disorders) | 0 | 0 | 20 | 14
Injury (Vascular disorders) | 0 | 0 | 1 | 0
Other (Vascular disorders) | 0 | 0 | 15 | 12
Pseudoaneurysm (Vascular disorders) | 0 | 0 | 2 | 3
Thrombosis/Thromboembolism (Vascular disorders) | 0 | 0 | 4 | 1
Thrombus (Vascular disorders) | 0 | 0 | 1 | 0
Retroperitoneal hematoma (Vascular disorders) | 0 | 0 | 0 | 1
MV surgery (Cardiac disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days